CLINICAL TRIAL: NCT02423889
Title: Stereotactic Radiotherapy in Low Risk Prostate Cancer: a Phase II Study
Brief Title: Stereotactic Volumetric Radiotherapy in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Stefano Vagge, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RITS13.001
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: Hypofractionated radiotherapy; SBRT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

ARMS (1):
- 1 (Experimental): Stereotactic radiotherapy with a total dose of 36.25 Gy in 5 fractions (7.25 Gy per fraction, 2 fractions per week) in low risk prostate cancer patients is delivered to evaluate acute and subacute toxicty
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy

SUMMARY:
This is a prospective, single arm, phase II, multicentric study. It evaluates the acute and late toxicity after stereotactic radiotherapy in low risk prostate cancer patients. All participants receive a total dose of 36.25 Gy in 5 fractions, twice a week, 7.25 Gy per fraction.

ELIGIBILITY:
Inclusion Criteria:

* Histology of prostate adenocarcinoma
* Age≥ 18 years
* Life expectancy≥ 10 years
* Clinical negative nodes (N0)
* No metastasis presence (M0)
* No previous pelvic radiation therapy
* Total PSA≤10 ng/ml
* Gleason score ≤ 6
* T1-2
* ≤ 3 positive biopsy at prostatic mapping
* Signed informed consent

Exclusion Criteria:

* Positive nodes (N+) or metastatic disease (M+)
* Inflammatory bowel disease, collagen- vascular disorders or active autoimmune disorders
* Anticoagulant treatment in progress
* Hip or pelvic presence of medical devices that could prevent a correct image acquisition
* Symptomatic haemorrhoidal disease
* Adverse reactions to iodinate or paramagnetic contrast media
* Previous malignant cancer, except basocellular skin tumour or other tumours healed since 5 years
* Previous pelvic radiotherapy
* Psychiatric disorder that preclude to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Acute toxicity | up to 3 months
  during treatment and up to 3 month from RT end
Late toxicity | up to 60 months
  since 4 month from RT end

SECONDARY OUTCOMES:
Disease free survival | up to 5 year
  Time from treatment end to biochemical recurrence or loco-regional recurrence or metastatic disease
Disease specific survival | up to 5 years
  Time from RT end to the date of patient death for cancer
Overall survival | up to 5 years
  Time from RT end to the date of patient death for any cause

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS AOU San Martino-IST, Genoa, GE
  - AO Città della salute e della scienza - Molinette, Turin, TO
  - Istituto del Radio "O. Alberti" Spedali Civili - University of Brescia, Brescia